CLINICAL TRIAL: NCT05924061
Title: The Role of Pentraxin 3 and Cathepsin B Levels in the Second Trimester in Predicting of Maternal and Fetal Results in Preeclamptic Pregnancy
Brief Title: The Role of Pentraxin 3 and Cathepsin B Levels in Preeclamptic Pregnancy
Status: Completed | Type: Observational
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor Department of Obstetrics and Gynecology, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Other Study IDs: 2011-KAEK-25 2021/09-09
Record Dates: First submitted 2023-04-04; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Pre-Eclampsia; Cathepsin B Level; Pentraxin 3 Level
Keywords: second trimester; preeclampsia; pentraxin 3; Cathepsin B
MeSH Terms: conditions — Pre-Eclampsia | interventions — Cathepsin B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women with preeclampsia between 20-28 weeks (study group): Maternal serum cathepsin B and pentraxin 3 levels in 20-28 weeks pregnant women with preeclampsia
  Interventions: Other: Cathepsin B and pentraxin 3 levels in preeclampsia with pregnant women
- Healthy pregnant women between 20-28 weeks ( control group): Maternal serum cathepsin B and pentraxin 3 levels in 20-28 weeks healthy pregnant women ( control group)
  Interventions: Other: Cathepsin B and pentraxin 3 levels in preeclampsia with pregnant women

INTERVENTIONS:
Other: Cathepsin B and pentraxin 3 levels in preeclampsia with pregnant women — The effect of cathepsin b and pentraxin 3 levels on maternal/fetal outcomes in pregnant women diagnosed with preeclampsia

SUMMARY:
In this study, the investigator aim was to compare Cathepsin B and Pentraxin 3 levels measured from maternal serum of pregnant women diagnosed with preeclampsia in the second trimester, the effects of these levels on maternal/ fetal outcomes and the composite results of Cathepsin B and Pentraxin 3 levels alone or together and contribute to the literature in this area.

DETAILED DESCRIPTION:
This prospective case-control study was conducted between 1 January 2022 and 31 December 2022 at Bursa Yuksek Ihtisas Training and Research Hospital. The study was conducted with pregnant women between ages of 18-45 who were diagnosed with preeclampsia in the second trimester. This study was conducted with total 156 pregnant women. participants were grouped according to the presence of preeclampsia; Group1: Patients diagnosed with preeclampsia between 20-28 weeks (study group) (n:78) , Group 2: Healthy pregnant women between 20-28 weeks without a diagnosis of preeclampsia ( control group) (n:78) . As soon as preeclampsia is diagnosed and before any treatment was started, maternal serum samples were collected in the Cathepsin B and Pentraxin 3 kit in amounts suitable for the study. The samples obtained were kept in biochemistry laboratory at -80 degrees until the study was conducted. After all samples were collected, Cathepsin B and Pentraxin 3 values were measured by ELISA method.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Pregnant women diagnosed with preeclampsia between 20-28 weeks of gestation
* Healthy pregnant women between 20-28 weeks of gestation who want to be involved in the study.

Exclusion Criteria:

* Multiple pregnancies
* Pregnant women who gave birth below 24 weeks of gestation
* Pregnant women diagnosed with other hypertensive diseases of pregnancy other than preeclampsia ( gestational hypertension, chronic hypertension, superimposed hypertension)
* Pregnant women with chromosomal or congenital anomalies in the fetus
* Women with a known infective or autoimmune disease before pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: singleton pregnancy white people socio-cultural differences were not considered
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the effects and composite results of cathepsin b and pentraxin 3 levels in pregnant women diagnosed with preeclampsia | 12 months
  serum cathepsin b (nmoL pNA/mL) and serum pentraxin 3 (ng/ml) levels composite results on pregnant women diagnosed with preeclampsia

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Nazlı YENIGUL, Bursa, Turkey (Türkiye)